CLINICAL TRIAL: NCT01757015
Title: A 26-week Multi-center Randomized Double-blind Study to Compare Efficacy and Safety of NVA237 Versus Placebo as an add-on to Maintenance Therapy With Fixed-dose Combination Salmeterol/Fluticasone Propionate in COPD Patients With Moderate to Severe Airflow Limitation
Brief Title: Safety and Efficacy of NVA237 as an add-on to Fixed Dose Combination LABA/ICS
Acronym: GLOW8
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237A2311; 2012-002854-21
Record Dates: First submitted 2012-12-17; First posted 2012-12-28 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2013-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Moderate to severe airflow limitation; GOLD spirometric classification 2 and 3; GOLD group B and D; NVA237; Salmeterol fluticasone propionate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo to NVA237 (50 μg) o.d. in the morning Patients will also receive open label salmeterol/fluticasone propionate (50/500 µg) b.i.d., in the morning and evening
  Interventions: Drug: Placebo to NVA237
- NVA237 (Experimental): NVA237 (50 μg) o.d. in the morning Patients will also receive open label salmeterol/fluticasone propionate (50/500 µg) b.i.d., in the morning and evening.
  Interventions: Drug: NVA237

INTERVENTIONS:
Drug: NVA237 — NVA237 (50µg, o.d. via SDDPI) in the morning,
  Arms: NVA237
Drug: Placebo to NVA237 — Placebo to NVA237
  Arms: Placebo

SUMMARY:
This study is to evaluate if add-on treatment with inhaled NVA237 (50 µg) once daily (o.d.) via single-dose dry-powder inhaler (SDDPI) further improves lung function and health status and is well tolerated compared to placebo in symptomatic COPD patients with moderate to severe airflow limitation who are already receiving maintenance therapy with inhaled fixed-dose-combination of salmeterol/fluticasone propionate (50/500 µg) twice daily (b.i.d.) via multi-dose dry powder inhaler (MDDPI).

ELIGIBILITY:
Inclusion Criteria:

* Current or ex-smokers who have a smoking history of at least 10 pack years (e.g., 10 pack years = 1 pack/day × 10 years, ½ pack/day × 20 years, etc.).
* COPD (Chronic Obstructive Pulmonary Disease) patients with moderate to severe airflow limitation (Spirometry classification: GOLD 2 or 3) at Visit 2:
* Post-bronchodilator FEV1 (Forced Expiratory Volume in one second) ≥30% and <60% of the predicted normal, and,
* Post-bronchodilator FEV1/forced vital capacity (FVC) <0.70
* Patients on maintenance treatment with fixed-dose combination of inhaled salmeterol and fluticasone propionate (50/500 µg) b.i.d. delivered via a proprietary MDDPI (multidose dry powder inhaler) device for at least 30 days prior to screening visit (Visit 1).
* Patients in category Gold B or D with a CAT (COPD Assessment Test) total score ≥10 at screening (Visit 1) and before randomization (Visit 3).
* Patients with a history of at least 1 moderate or severe COPD exacerbation within the previous year.

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of child-bearing potential, unless they are using effective methods of contraception during the study
* Patients with a history of long QT syndrome or whose QTc measured at run-in (Visit 2) (Fridericia method) is prolonged (>450 ms). (These patients cannot be re-screened.)
* Patients with evidence (upon visual inspection) of oropharyngeal candidiasis at baseline with or without treatment.
* Patients who have not achieved an acceptable spirometry result at run-in (Visit 2) in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria for acceptability and repeatability.
* Patients who have had a COPD exacerbation that required treatment with antibiotics or oral corticosteroids or hospitalization in the 6 weeks prior to screening (Visit 1).
* Patients who have had a respiratory tract infection within 4 weeks prior to screening (Visit 1).
* Patients requiring long term oxygen therapy prescribed for >12 hours per day.
* Patients with allergic rhinitis who use an H1 antagonist or intra-nasal corticosteroids intermittently. (Treatment with a stable dose or regimen is permitted.)
* Patients with concomitant pulmonary disease (e.g., lung fibrosis, sarcoidosis, interstitial lung disease, or pulmonary hypertension), clinically significant bronchiectasis, or history of pulmonary lobectomy, lung volume reduction surgery, or lung transplantation.
* Patients with active pulmonary tuberculosis, unless confirmed by imaging to be no longer active.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Trough Forced Expiratory Volume in 1 second (FEV1) | after 12 weeks of treatment
  Comparison of NVA237 treatment versus placebo treatment in the trough FEV1 after 12 weeks of treatment

SECONDARY OUTCOMES:
Total score of St George's Respiratory Questionnaire for COPD patients (SGRQ-C). | 26 weeks
  Comparison of NVA237 treatment versus placebo treatment in terms of change in SGRQ-C after 26 weeks of treatment
Trough Forced Expiratory Volume in 1 second (FEV1) | week 4 , week 26
  Comparison of effect of NVA237 treatment versus placebo treatment in FEV1 after 4 weeks and after 26 weeks of treatment
Total score of the Transition Dyspnea Index (TDI) | Week 12 and week 26
  Comparison of effect of NVA237 treatment versus placebo treatment in the total TDI score after 12 weeks and after 26 weeks of treatment
Assessment of safety and tolerability | 26 Weeks
  All safety endpoints will be summarized for the safety set.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals